CLINICAL TRIAL: NCT03921788
Title: Study of the Role of Vasoactive Neuropeptides in the Genesis of Venous Pelvic Pain
Brief Title: Neuropeptides and Venous Pelvic Pain
Acronym: NVPP
Status: Completed | Type: Observational
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Sergey Gavrilov, MD, PhD, Professor of the Department of Faculty Surgery №1, Pirogov Russian National Research Medical University
Other Study IDs: 01201254811
Record Dates: First submitted 2019-04-12; First posted 2019-04-19 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Pelvic Pain; Varicose Veins Pelvic; Pelvic Congestion Syndrome
Keywords: venous pelvic pain; pelvic congestion syndrome; calcitonin gene-related peptide; substance P
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Patients with venous pelvic pain. Pain measurement using a visual analogue scale, the study of calcitonin gene-related peptide and substance P (ELISA)
- Group 2: Patients without venous pelvic pain. Pain measurement using a visual analogue scale, the study of calcitonin gene-related peptide and substance P (ELISA)
- Group 3: Volunteers without pain syndromes of any location. Pain measurement using a visual analogue scale, the study of calcitonin gene-related peptide and substance P (ELISA)

SUMMARY:
Mechanisms of the development of pain in chronic venous diseases (CVD), including pelvic congestion syndrome (PCS), are studied incompletely. The existing hypotheses of the occurrence of venous pelvic pain (VVP) do not allow to answer the question why some patients have no pain syndrome while others have very pronounced pain despite the same morphofunctional changes in the pelvic veins? The investigators are planning to carry out a study aimed at studying the content of calcitonin gene-related peptide (CGRP) and substance P (SP) in the serum of patients with pelvic veins and pelvic pain, and to study the relationship between the values of CGRP and SP in these patients.

DETAILED DESCRIPTION:
The first phase of the study includes a set of 3 patient groups: the first is patients with pelvic vein dilation and blood reflux through them in combination with venous pelvic pain; the second is patients with pelvic vein dilatation without venous pelvic pain. The third, control group will include healthy female volunteers without pelvic veins and any chronic pain syndromes.

At the second stage of the study, a study will be made of the levels of calcitonin gene-related peptide (CGRP) and the substance P (SP) in the serum using an ELISA method. In addition, after studying the content of the CGRP and SP in the serum of volunteers, the investigators expect to obtain the reference values of these neuropeptides. In this phase of the study, a statistical analysis of the data obtained will be carried out, a correlation analysis between venous pelvic pain and the level of the CGRP and CP.

The data for each patient will be entered into a specially designed patient questionnaire. It will include clinical and ultrasound data, results of ELISA.

ELIGIBILITY:
Inclusion Criteria:

* The reproductive age of the woman
* Blood reflux in the parametric, uterine, gonadal veins
* The absence of any concomitant pathology, accompanied by chronic pelvic pain

Exclusion Criteria:

* The absence of blood reflux in in the parametric, uterine, gonadal veins
* The presence of diseases, the clinical course of which suggests the presence of chronic pelvic pain and other varieties of chronic pain, including migraine
* Pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women aged 18-45 years
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
The severity of venous pelvic pain | 5 min
  For the quantitative determination of the severity of venous pelvic pain using a visual analogue scale, measurement in points. The visual analogue scale (VAS) consists of a straight line with the endpoints defining extreme limits such as "no pain at all" and "pain as bad as it could be". The patient is asked to mark his pain level on the line between the two endpoints. The distance between "no pain at all" and the mark then defines the subject's pain.
The level of calcitonin-gene-related peptide | 22 hours
  Protocol V (Ab1hr.Std2hr. BtON) was used for the enzyme-linked immunosorbent assay (ELISA).
  The indicator is measured in ng / ml
The level of substance P | 22 hours
  Protocol V (Ab1hr.Std2hr. BtON) was used for the enzyme-linked immunosorbent assay (ELISA).
  The indicator is measured in ng / ml

CONTACTS AND LOCATIONS:
Overall Officials: Natalia V Koroleva, PhD, Study Chair — Pirogov Russian National Research Medical University
Locations (1):
- Department of Faculty Surgery №1, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] FitzGerald MP. Chronic pelvic pain. Curr Womens Health Rep. 2003 Aug;3(4):327-33. PMID 12844458
- [Result] Stones RW, Thomas DC, Beard RW. Suprasensitivity to calcitonin gene-related peptide but not vasoactive intestinal peptide in women with chronic pelvic pain. Clin Auton Res. 1992 Oct;2(5):343-8. doi: 10.1007/BF01824305. PMID 1422102
- [Result] Origoni M, Leone Roberti Maggiore U, Salvatore S, Candiani M. Neurobiological mechanisms of pelvic pain. Biomed Res Int. 2014;2014:903848. doi: 10.1155/2014/903848. Epub 2014 Jul 8. PMID 25110704